CLINICAL TRIAL: NCT04220190
Title: Phase 2/3 Trial of Autologous Hybrid TREG/Th2 (RAPA-501) T Stem Cell Therapy for Amyotrophic Lateral Sclerosis
Brief Title: RAPA-501 Therapy for ALS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rapa Therapeutics LLC (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPA-501-ALS
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; RAPA-501; Autologous TREG/Th2 T stem cell therapy; Orphan Disease; rare disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Rare Diseases

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RAPA-501 Autologous T stem cells (Experimental): Phase 2/3 Expansion Cohort, Single-agent RAPA-501 T stem cells 80 x 10EE6 cells per infusion (no host conditioning)
  Interventions: Biological: RAPA-501 Autologous T stem cells

INTERVENTIONS:
Biological: RAPA-501 Autologous T stem cells — Experimental: Phase 2/3 Expansion Cohort, Single-agent RAPA-501 T stem cells 80 x 10EE6 cells per infusion (no host conditioning)
  Other Names: RAPA-501 cells

SUMMARY:
RAPA-501-ALS is a phase 2/3 expansion cohort study of RAPA-501 autologous hybrid TREG/Th2 cells in patients living with amyotrophic lateral sclerosis (pwALS).

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center phase 2/3 study evaluating RAPA-501 T stem cell therapy in pwALS on an expansion cohort. Amyotrophic lateral sclerosis (ALS) is a rare disease that is also considered an orphan disease according to the Orphan Drug Act.

After a subject consents to the study, an apheresis procedure will be performed to collect cells to manufacture the investigational product, RAPA-501 T stem cells. RAPA-501 T stem cells are manufactured ex vivo using epigenetic reprogramming to yield a T stem cell population that is enriched for a dual anti-inflammatory phenotype based on hybrid TREG and Th2 differentiation. RAPA-501 cells express both the TREG and Th2 transcription factors FOXP3 and GATA3, are enriched for expression of the ATP ectonucleotidase molecules CD39 and CD73, are enriched for the T cell homing molecule CD103, and suppress both effector T cell inflammatory molecules and CNS microglial cell inflammatory molecules.

This study consists of a phase 2/3 expansion cohort that is evaluating RAPA-501 T stem cell therapy at the dose of 80 x 10EE6 cells per infusion, with up to 4 infusions separated by six weeks between doses (infusion at time 0, and then after week 6, 12, and 18). Study subjects are then followed at the treatment site at 24 weeks and 30 weeks on-study; then, subjects are followed remotely using surveys for two years to capture major clinical events and assess survival. The primary objective in the expansion cohort is to determine the feasibility and safety of the highest established safe dose of RAPA-501 (80 x 10EE6 cells per infusion) in patients with standard-risk ALS (as defining by study entry values of: SVC greater than or equal to 70% of predicted normal; time interval since first ALS symptom, 24 months or less; and ALSFRS-R score between 34 and 45). Secondary study objectives relate to assessing the potential efficacy of RAPA-501 therapy through monitoring of ALSFRS-R scores, SVC values, time to King's stage transition, and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Patients with sporadic or familial amyotrophic lateral sclerosis (ALS) diagnosed as laboratory-supported possible, probable, or definite according to World Federation of Neurology El Escorial Criteria.
3. . Less than or equal to 24 months since ALS symptom onset.
4. Total ALSFRS-R score between 34 and 45.
5. Must have a source of autologous T cells potentially sufficient to manufacture RAPA-501 cells, as defined by a peripheral CD3+ T cell count ≥ 500 cells per μl.
6. Patients may continue riluzole (Rilutek®), and/or edaravone (Radicava®), and/or sodium phenylbutyrate/taurusodial (Relyvrio™) if on a stable dose for at least 30 days prior to the screening visit.
7. Patients must be ≥ 2 two weeks removed from major surgery or investigational therapy.
8. Patients must have recovered from clinical toxicities ([resolution of CTCAE(v5) [version 5] toxicity to a value of ≤ 2].).
9. Serum creatinine ≤ less than or equal to 2.0 mg/dL.
10. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN).
11. Bilirubin ≤ 1.5 (except if due to Gilbert's disease).
12. Pulmonary slow vital capacity (SVC) ≥ 70% of predicted normal.
13. No history of abnormal bleeding tendency.
14. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Active uncontrolled infection.
2. Hypertension not adequately controlled by ≤ 3 medications.
3. History of documented pulmonary embolus within 6 months of enrollment.
4. Clinically significant cardiac pathology, as defined by: myocardial infarction within 6 months prior to enrollment, Class III or IV heart failure according to NYHA, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
5. Patients with history of coronary artery bypass grafting or angioplasty will receive a cardiology evaluation and be considered on a case-by-case basis.
6. HIV, hepatitis B, or hepatitis C seropositive.
7. Pregnancy or breastfeeding patients.
8. Patients of Subjects of childbearing age, or males who have a partner of childbearing potential, who are unwilling to practice contraception.
9. Patients Subjects may be excluded at the Principal Investigator discretion of the PI or if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
In the expansion cohort enrolling standard-risk pwALS, determine the feasibility and safety of the highest established safe dose of RAPA-501 (80 x 10^6 cells per infusion). | Through 30 Weeks On-Study

SECONDARY OUTCOMES:
Characterize immune system parameters pre- and post-therapy. | Through 30 Weeks On-Study
  Specifically, relative to pretreatment patient peripheral blood values, determine whether study interventions: (a) increase circulating Th2 and TREG cells; (b) reduce circulating Th1 cells; (c) increase T cell expression of programmed death-1 (PD-1); and (d) reduce inflammatory cytokines IL-1-beta, IL-6, and TNF-alpha.
Relative to pretreatment values, characterize the potential effect of RAPA-501 therapy on serum markers of neurodegeneration (neurofilament light, NfL). | Through 30 Weeks On-Study
Relative to pretreatment values, characterize the potential effect of RAPA-501 therapy on pulmonary function, as measured by slow vital capacity measurements (SVC, percent of predicted normal). | Through 30 Weeks On-Study
Relative to pretreatment values, characterize the potential effect of RAPA-501 therapy on hand grip strength using hand-held dynamometry. | Through 30 Weeks On-Study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fowler, M.D., Study Director — Rapa Therapeutics LLC
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No